CLINICAL TRIAL: NCT00141674
Title: A Prospective Randomized Controlled Trial Comparing the Effects of Fresh vs. Old Blood on Cerebral Oxygen Extraction in Patients With Traumatic Brain Injuries
Brief Title: Age of Blood in Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Dean Chittock, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C04-0459; VCHRI #V04-0261
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Traumatic Brain Injury
Keywords: Blood transfusion; Age of blood; Traumatic Brain Injury; Cerebral Oxygen Extraction Ratio; Age of transfused blood in traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Procedure: Blood Transfusion — This is a single centre randomized trial in severely head injured patients requiring a blood transfusion. Randomization will be by computer generated random numbers paced in sealed envelopes. Patients would be randomized to receive either blood less than 5 days old or greater than 20 days old. The decision to transfuse and all other intensive care management will be unaltered by enrolment in the study.

SUMMARY:
Donated red blood cells vary in how old they are, that is, how long they have been stored since being collected from donors. Blood that has been donated is stored for a maximum of 42 days, after this time it is expired. That means that red blood cells that are given to patients as a blood transfusion can be anywhere from a few days old to 42 days old. The average age of blood that is given as a blood transfusion in this hospital is 21 days old.

As stored blood gets older its ability to carry oxygen may be reduced. Whether or not this is important in patients with a brain injury is not currently known.

The purpose of this study is to try and determine if fresh blood (less than 5 days old) is better than old blood (greater than 20 days old) in improving the supply of oxygen in patients who have suffered an injury to their brain.

DETAILED DESCRIPTION:
PURPOSE

To demonstrate that packed red blood cells (pRBC) less than 5 days old are superior to older (>20days) blood in improving markers of cerebral oxygenation in acutely head injured patients.

HYPOTHESIS

Transfusion of pRBC will result in increased cerebral extraction of oxygen. This effect will be greatest in pRBC stored for a greater length of time.

JUSTIFICATION

One of the main aims of the intensive management of head injured patients is the prevention of secondary hypoxic or hypotensive insults in the already injured brain. Packed red blood cell transfusions are commonly given to trauma patients suffering anemia (Hgb <100 g/l) secondary to blood loss in order to improve oxygen delivery to vital organs including the brain.

Previous studies have shown that the capacity of packed red blood cells (pRBC) to improve oxygen delivery to tissues diminishes with increased time in storage. This storage lesion may improve with time post transfusion; however, this may take many hours.

Other studies have shown an association between age of pRBCs transfused and length of stay in trauma patients and mortality in septic ICU patients. Unused old blood is likely to be sent to high volume centers to avoid wasting a precious resource.

The effects of 'old' transfused blood have not been subject to rigorous prospective studies and age of blood has not been shown to be causally related to the adverse outcomes mentioned above, hence the need for further studies.

The injured brain is uniquely sensitive to further damage. Even a brief secondary insult of either hypotension or hypoxia has been shown to have a significant adverse effect on outcomes including permanent disability and death. Furthermore the measurement of markers of cerebral oxygenation forms part of the standard care of severely head injured patients in this institution giving a unique opportunity to study the effects of blood transfusion in this group of patients.

The presence of a storage lesion in pRBCs lasting even a few hours could have a significant impact on the head injured patient. If indeed 'fresh' blood does significantly improve markers of cerebral oxygenation when compared to older blood it could alter clinical practice significantly by placing a priority on transfusing only 'fresh' blood in such patients. The effect of age of pRBCs has never been studied in the head injured population.

Donated blood is stored for a maximum of 42 days. The average age of pRBC administered at VGH is 21 days.

OBJECTIVES

To evaluate the effect of transfusing "fresh" (blood stored less than 5 days) versus "stored" (blood stored for greater than 20 days) pRBC on cerebral oxygen extraction. We will also evaluate the effect of transfusion of pRBC on cerebral oxygen extraction in patients with traumatic brain injury.

RESEARCH METHOD

This is a single centre randomized trial in severely head injured patients requiring a blood transfusion. Randomization will be by computer generated random numbers paced in sealed envelopes. Patients would be randomized to receive either blood less than 5 days old or greater than 20 days old. The decision to transfuse and all other intensive care management will be unaltered by enrolment in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary traumatic brain injury
2. Glasgow Coma Scale < 8
3. Invasive neurological monitoring:

   1. External Ventricular Drain
   2. Jugular bulb catheter
4. Hemoglobin < 100 g/L and decision has been made by Attending Physician to treat with one unit pRBC

Exclusion Criteria:

1. Age < 16
2. Ongoing need for blood products
3. Received Packed Red Blood Cells within preceding 24 hours
4. Multiple trauma necessitating ongoing resuscitation
5. Pregnant patients
6. Chronic renal failure
7. Severe sepsis or septic shock
8. Adult respiratory distress syndrome or acute lung injury
9. Presumed unstable neurological status during course of study
10. Lack of informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of transfusing "fresh" (blood stored less than 5 days) versus "stored" (blood stored for greater than 20 days) packed red blood cells (pRBC) on cerebral oxygen extraction ratio for 24 hours post transfusion | 20 days

SECONDARY OUTCOMES:
To evaluate the effect of transfusion of pRBC on cerebral oxygen extraction in patients with traumatic brain injury for 24 hours post transfusion. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dean Chittock, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada